

Final 1.0/ 21-Dec-2023

# **SPONSOR:**

# **Autolus**

# **PROTOCOL NUMBER:**

AUTO3-DB1

# STATISTICAL ANALYSIS PLAN

| Author: | |
|----------|-------------|
| Version: | Final 1.0 |
| Date: | 21-Dec-2023 |



Final 1.0/ 21-Dec-2023

# 1 Cover and signature pages

| Sponsor: | Autolus |
|---|---|
| Protocol Number: | AUTO3-DB1 |
| Study Title: | A Single-arm, Open-label, Multi-centre, Phase I/II Study Evaluating the Safety and Clinical Activity of AUTO3, a CAR T Cell Treatment Targeting CD19 and CD22 with Anti PD-1 Antibody in Patients with Relapsed or Refractory Diffuse Large B Cell Lymphoma |
| Document Version No | Final 1.0 |

We, the undersigned, confirm that we have read, understood and agree to the content of this document and hereby authorize its approval.

| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
|------|------------------------------------------------|-------|-----------|
| | Senior Biostatistici | an II | |



Final 1.0/ 21-Dec-2023

| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
|------|------------------------------------------------|------|-----------|
| | Director | | |

| Name | Title<br>[text box when using<br>eSignatures]: | Date | Signature |
|---|---|---|---|
| | VP, Head of Clinica | al Developmen | <u> </u> |



Protocol: AUTO3-DB1

# **Statistical Analysis Plan:**

Final 1.0/ 21-Dec-2023

# **Table of Contents**

| 1 | Cove | er and signature pages | . 2 |
|---|-------|------------------------------------------------------------|-----|
| 2 | List | of Abbreviations and Definition of Terms | 6 |
| 3 | Intro | oduction | 9 |
| 4 | Stud | ly Objectives | 9 |
| 5 | Stud | ly Design | |
| | 5.1 | STUDY DESIGN AND POPULATION | 11 |
| | 5.2 | STUDY TREATMENTS AND ASSESSMENTS | 13 |
| | 5.3 | RANDOMISATION AND BLINDING | 17 |
| | 5.4 | SAMPLE SIZE JUSTIFICATION | 18 |
| 6 | Stati | istical Considerations | |
| | 6.1 | TERMINATION OF THE STUDY AFTER END OF PHASE I | 19 |
| | 6.2 | SOFTWARE | |
| | 6.3 | MISSING DATA HANDLING | 19 |
| | 6.4 | PARTIAL DATE IMPUTATION | 19 |
| | 6.5 | VISIT WINDOWING | 23 |
| | 6.6 | BASELINE | 23 |
| | 6.7 | REPORTING GUIDELINES | 23 |
| 7 | Anal | lysis Sets | 28 |
| | 7.1 | ANALYSIS SETS | |
| | 7.2 | PROTOCOL DEVIATIONS | |
| 8 | Met | hods of Analyses and Presentations | |
| | 8.1 | PATIENT DISPOSITION | |
| | 8.2 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | |
| | 8.3 | PRIOR LYMPHOMA THERAPIES | |
| | 8.4 | MEDICAL HISTORY | |
| | 8.5 | PRIOR AND CONCOMITANT MEDICATIONS | |
| | 8.6 | BRIDGING THERAPIES AND NEW ANTI-CANCER THERAPIES | |
| | 8.7 | IMMUNOGLOBULIN THERAPIES | 31 |
| | 8.8 | LEUKAPHERESIS | |
| | 8.9 | LYMPHOMA B-SYMPTOMS | |
| | 8.10 | STUDY TREATMENT | |
| | 8.11 | FOLLOW-UP TIMES | |
| | 8.12 | EFFICACY DATA ENDPOINTS AND ANALYSES | |
| | 8.12 | 1 Primary Efficacy Endpoint and Analyses | |
| | 8.12 | , , , , | |
| | 8.12 | , , , , | |
| | 8.12 | , | |
| | 8.12 | | |
| | 8.13 | PHARMACODYNAMIC AND PHARMACOKINETIC ENDPOINTS AND ANALYSES | |
| | 8.14 | QUALITY OF LIFE OR PHARMACOECONOMIC ENDPOINTS AND ANALYSES | 37 |
| | 8.15 | SAFETY DATA ENDPOINTS AND ANALYSES | 37 |



# Protocol: AUTO3-DB1

# **Statistical Analysis Plan:**

# Final 1.0/ 21-Dec-2023

| | 8.15.1 | L Adverse Events (AEs) | 37 |
|---|---|---|---|
| | 8.15.2 | 2 Clinical Laboratory Evaluations | 39 |
| | 8.15.3 | 3 12-lead Electrocardiogram (ECG) | 39 |
| | 8.15.4 | Echocardiogram (ECHO) or Multiple Gated Acquisition (MUGA) | 39 |
| | 8.15.5 | 5 Vital Signs | 40 |
| | 8.15.6 | Physical and Neurological Examination | 40 |
| | 8.15.7 | 7 Eastern Cooperative Oncology Group (ECOG) Performance Status | 40 |
| | 8.15.8 | B Death information | 40 |
| | 8.15.9 | 9 Hospitalisation information | 41 |
| | 8.15.2 | | 41 |
| 9 | Interi | m Analyses | 41 |
| 10 | Devel | opment safety update report | 41 |
| 11 | Chan | ges to Planned Analyses | 41 |
| 12 | Docui | ment History | 42 |
| 13 | | ences | |
| 14 | Appe | ndices | 43 |
| 1 | L4.1 A | APPENDIX A – Study assessments | 43 |
| 1 | L4.2 | APPENDIX B – Lugano Classification (Cheson et.al 2014) | 43 |
| 1 | L4.3 A | APPENDIX C – Clinical Laboratory Tests Performed by Local Laboratory | 48 |
| 1 | 14.4 | Fables, Figures and Listing shells | 49 |



Final 1.0/ 21-Dec-2023

# 2 List of Abbreviations and Definition of Terms

AE Adverse Event

AESI Adverse Event of special interest

ALT Alanine Aminotransferase

ATC Anatomical Therapeutic Chemical

ASCT Autologous haematopoietic stem cell transplantation
ATIMP Advanced therapy investigational medicinal product

BM Bone marrow

BOR Best overall response

CAR Chimeric antigen receptor CD Cluster of differentiation

CDISC Clinical Data Interchange Standards Consortium

CI Confidence interval
CR Complete response
CRF Case Report Form

CRS Cytokine release syndrome

CSF Cerebrospinal fluid

CT Computed tomography

CTCAE Common Terminology Criteria for Adverse Events

CY Cyclophosphamide

DLBCL Diffuse large B cell lymphoma

DNA Deoxyribonucleic acid
DLT Dose limiting toxicity
DOR Duration of response

DSUR Development safety update report

ECG Electrocardiogram
ECHO Echocardiogram

ECOG Eastern Cooperative Oncology Group

eCRF Electronic Case Report Form

FDG Fluorodeoxyglucose

FISH Fluorescence In Situ Hybridization

Template Author: Version 5.0 25Jun2020


BMSOP111/F2



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

FL Follicular lymphoma

FLU Fludarabine

FLU-CY Fludarabine and Cyclophosphamide

GI Gastrointestinal

HIV Human immunodeficiency virus

i.v. Intravenous(ly)

ICAN Immune effector cell-associated neurotoxicity syndrome

ICH International Conference on Harmonisation

IFN Interferon

Ig Immunoglobulin

IHC Immunohistochemistry

IPI International prognostic index IVIG Intravenous immunoglobulin

LDH Lactate dehydrogenase

LVEF Left ventricular ejection fraction

MedDRA Medical Dictionary for Regulatory Activities

MRI Magnetic resonance imaging
MTD Maximum Tolerated Dose
NCI National Cancer Institute

NE Not evaluable

NT Neurotoxicity

OS Overall survival

PBMCs Peripheral blood mononuclear cells

PCR Polymerase chain reaction

PD Progressive Disease

PD-1 Programmed cell death protein 1

PD-L1 Programmed cell death ligand 1

PDvs Protocol deviations

PET Positron emission tomography

PFS Progression-free survival

PR Partial Response
PT Preferred Term

Template Author: Version 5.0 25Jun2020




Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

Q1 25% quartile Q3 75% quartile

qPCR Quantitative polymerase chain reaction

QTCF Heart rate-corrected QT interval (Fridericia's formula)

RCR Replication competent retrovirus

RP2D Recommended Phase II dose

SAE Serious adverse event
SAP Statistical analysis plan
SCT Stem cell transplant

SD Stable Disease

SD Standard deviation

SEC Safety Evaluation Committee

SI International System
SOC System Organ Class

TNF Tumour necrosis factor

TEAE Treatment-emergent adverse event

TFL(s) Table(s), Figure(s), Listing(s)

WBC White blood cell

WHODDE World Health Organization drug dictionary



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

# 3 Introduction

The purpose of this document is to describe the statistical methods, data derivations and data summaries to be employed in the analysis of study AUTO3-DB1 for Autolus in AUTO3, a chimeric antigen receptor (CAR) T cell treatment targeting cluster of differentiation (CD) 19 and/or CD22 followed by consolidation with anti-programmed cell death protein 1 (PD-1) antibody in subjects with relapsed or refractory diffuse large B Cell lymphoma (DLBCL).

The preparation of this statistical analysis plan (SAP) has been based on International Conference on Harmonisation (ICH) E3 and E9 Guidelines, in reference to Protocol AUTO3-DB1 Version 10.0 (06-May-2021) and latest available aCRF (14-Dec-2022).

# 4 Study Objectives

# **PRIMARY OBJECTIVES**

The primary objectives of the study are defined on Phase I and Phase II as follows:

- Primary objectives for Phase I:
  - Escalation:
    - To assess the safety and tolerability of AUTO3 administration with pembrolizumab;
    - To identify the recommended Phase II doses (RP2D) and maximum tolerated dose (MTD), if an MTD exists, of AUTO3.
  - Expansion:
    - To assess the safety and tolerability of AUTO3 administration with pembrolizumab in the outpatient/ambulatory care setting.
- Primary objectives for Phase II:
  - To evaluate the clinical efficacy of AUTO3 at the RP2D(s) with pembrolizumab in Cohort 1;
  - To assess the overall safety and tolerability of AUTO3 with pembrolizumab in Cohort 2 at the RP2D(s).

Template Author:
Version 5.0 25Jun2020


BMSOP111/F2



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

# **SECONDARY OBJECTIVES**

- To assess the overall safety and tolerability of AUTO3 with pembrolizumab;
- To evaluate the feasibility of generating the advanced therapy investigational medicinal product (ATIMP), AUTO3;
- To evaluate the overall clinical efficacy of AUTO3 with pembrolizumab;
- To determine the expansion and persistence of AUTO3 following adoptive transfer in different lymphoma subtypes;
- Duration of B-cell aplasia.

# **EXPLORATORY OBJECTIVES**

- To determine the time course and magnitude of cytokine release evaluated using an appropriate assay;
- To evaluate the effect of anti-PD-1 antibody on the time course and magnitude of cytokine release using an appropriate assay;
- To assess the duration of depletion of circulating B cells as determined by flow cytometry on the peripheral blood and correlate this with disease response;
- To assess antibody and/or T cell mediated immune responses against AUTO3;
- To characterise the relationship between the CAR T cell phenotype/genomics and persistence *in vivo*;
- Seek any relationship between parameters of activity, level of CD19 or CD22 expression (flow cytometry), tumour programmed cell death ligand 1 (PD-L1) expression, and CAR T cell phenotype;
- Seek any relationship between incidence and severity of cytokine release syndrome (CRS), neurotoxicity (NT) or other toxicity, and tumour burden, level of CD19 or CD22 expression [immunohistochemistry (IHC) or flow cytometry], CAR T cell phenotype, and PD-1 expression;
- To evaluate cerebrospinal fluid (CSF) for potential markers associated with NT.



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

# 5 Study Design

# 5.1 STUDY DESIGN AND POPULATION

The study patient population for this study is DLBCL and large B cell lymphoma subsets, and will include:

- DLBCL, not otherwise specified (NOS), per World Health Organisation classification and DLBCL with MYC and BCL2 and/or BCL6 rearrangements (double/triple hit);
- Transformed DLBCL from follicular lymphoma (FL);
- Transformed DLBCL from other indolent lymphomas (excluding Richter's transformation);
- High-grade B cell lymphoma with MYC expression (excluding Burkitt's lymphoma);
- Primary mediastinal large B cell lymphoma.

In addition, since this is an experimental therapy, the study patient population will be restricted to patients with chemotherapy-refractory disease, or relapse after at least two lines of therapy (including an anti-CD20 monoclonal antibody (unless tumour is CD20-negative) and an anthracycline cycle), or after autologous haematopoietic stem cell transplantation (ASCT) and have PET positive disease (for efficacy assessment).

The study is a single-arm, open-label, multi-center, Phase I/II dose-escalation and expansion study, evaluating the safety and clinical activity of AUTO3 with anti-PD-1 antibody (pembrolizumab) when administered to patients with confirmed diagnosis of relapsed or refractory DLBCL and large B cell lymphoma subsets. The study will consist of 2 parts, a Phase I (dose escalation) followed by a Phase II (dose expansion).

#### Phase I

Dose escalation: To identify the optimal dose (based on safety, tolerability, and anti-tumour activity) of AUTO3 using a rolling 6 dose escalation design. Up to 4 cohorts and approximately 30 patients with DLBCL (and its defined subsets) will be enrolled. Each cohort dose may include up to 6 patients, except Cohort 1 which may include up to 12 patients (3 patients without consolidation therapy, and 3-6 patients with consolidation therapy). Doses from 50 × 10<sup>6</sup> to 900 × 10<sup>6</sup>



Final 1.0/ 21-Dec-2023

CD19/CD22 CAR-positive T cells, administered as a single dose will be evaluated. All patients (except the first three patients in the dose level 1 cohort) will receive limited consolidation or pre-conditioning therapy with pembrolizumab.

- Expansion cohort: To assess the safety and tolerability of AUTO3 at the recommended phase 2 dose(s) (RP2Ds) or dose range and pembrolizumab regimen identified in the dose escalation part. Approximately 20 patients with DLBCL will be treated in an outpatient/ambulatory care setting.
- Phase II: To further characterise the safety and assess the efficacy and anti-tumour activity of AUTO3 at the recommended dose(s) or dose range schedule confirmed in Phase I; approximately up to 101 patients will be treated in the dose expansion phase (81 patients with DLBCL subsets and transformed follicular lymphoma in Cohort 1 and, additionally, 20 patients in Cohort 2 with primary mediastinal large B cell lymphoma and those with lymphoma transformed from other indolent histologies).

Approximately up to 171 patients in total are expected to be enrolled (consented) into Phase I and Phase II of the study and approximately 151 patients in total are anticipated to be treated with AUTO3 therapy.

An overview of the study design is presented in <u>Figure 1</u> below.

Figure 1. Dose Escalation and Dose Expansions Phases



The total study duration is estimated to approximately 7 years from first patient enrolled to the end of study. The end of the study is defined as the last patient last visit (LPLV), expected to be



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

36 months after the last patient's AUTO3 dose or earlier in the event of patient death or consent withdrawal.

In the event of disease progression prior to the end of the study, patients will continue to be monitored for safety and survival in order to collect Health Authority requested data (e.g. delayed AEs) until the end of the study or until time of early withdrawal or death. The survival follow-up can be conducted via telephone contact if necessary.

At the end of the study or following AUTO3 treatment and early withdrawal from this study, all patients will be followed until death or withdrawal of consent for up to 15 years following their last AUTO3 infusion under a separate long-term follow-up study protocol.

# **5.2 STUDY TREATMENTS AND ASSESSMENTS**

The study will consist of the following six stages:

- **Screening**: After providing written informed consent for study participation, all patients will be screened for study eligibility. Eligible patients will proceed to leukapheresis.
- Leukapheresis: Eligible patients will undergo leukapheresis to facilitate manufacture of the ATIMP, AUTO3. Once leukaphereses is accepted for manufacturing, the patient will be enrolled on the study.
- Pre-Conditioning: If sufficient AUTO3 is successfully manufactured and released, and
  the patients continue to meet eligibility requirements for the study, they will proceed to
  receive a standard lymphodepleting pre-conditioning treatment with fludarabine (FLU)
  for 4 days and cyclophosphamide (CY) for 2 days, to end 3 days before AUTO3 infusion.
  For Regimen B, pre-conditioning will include in addition to FLU and CY a single dose of
  pembrolizumab, 200 mg given on Day -1.
- Treatment: AUTO3 will be administered intravenously (i.v.) as a single infusion on Day 0. The treatment phase will extend from Day 0 (infusion day) until Day 28 post AUTO3 administration. Patients are expected to be monitored closely (in hospital or ambulatory care as clinically appropriate) for 10 days or longer if clinically necessary for monitoring and management.
- Consolidation: Provided any acute toxicities have resolved, anti-PD1 antibody



Final 1.0/ 21-Dec-2023

(pembrolizumab, 200 mg infused over 30 min) will be administered for Regimen A on Days 14, 35 and 56 (±3 days).

• **Follow-up**: The follow-up phase will begin 1 month post AUTO3 infusion and at end of the study; at death or withdrawal of consent, which ever happens first.

An overview of the six study stages is presented in Figure 2.

Figure 2. Overview of the Stages of the Study





From signing of consent until the End of Study visit, information relating to AEs, laboratory abnormalities, disease response and biomarker changes will be collected according to the AE reporting period. The schedule of assessments to be performed during the study is detailed in Appendix A.

Eligible patients will receive a single dose i.v. infusion of AUTO3 following pre-conditioning



Final 1.0/ 21-Dec-2023

treatment. The AUTO3 product contains both transduced (CD19/CD22 CAR-positive) and non-transduced T cells. The dose is expressed as the number of CD19/CD22 CAR-positive T cells. Below dose levels are planned in Phase I:

- Dose Level 1: 50 x 10<sup>6</sup> CD19/CD22 CAR-positive T cells;
- Dose Level 2: 150 x 10<sup>6</sup> CD19/CD22 CAR-positive T cells;
- Dose Level 3: 450 x 10<sup>6</sup> CD19/CD22 CAR-positive T cells;
- Dose Level 4: 900 x 10<sup>6</sup> CD19/CD22 CAR-positive T cells.

The treatment phase will involve infusion of AUTO3 on Day 0. Patients will be monitored for up to 10 days (inpatient or ambulatory care setting), or longer if clinically necessary.

During Phase I the Safety Evaluation Committee (SEC) will meet after the first patient in every cohort completes 14 days, to confirm continuation of enrolment to that cohort and thereafter meet again after the third and or sixth patient in a cohort has completed the dose limiting toxicity (DLT) assessment period. Only after a cohort is declared safe by the SEC can the next higher dose level be opened. Back filling of a cohort (maximum n=6 evaluable patients /cohort) declared safe may be undertaken in parallel to the ongoing enrolment of a higher dose level, to obtain additional biomarker and safety data. All patients will be evaluated for efficacy. A minimum dosing interval of 7 days will be maintained between patients even if they are enrolled to a cohort that is declared safe in the Phase I part of the study.

The planned study cohorts for Phase I are presented in Table 1.

Table 1: Study Treatment Cohorts (phase I/dose escalation)

| Dose<br>Levels | Treatment<br>Cohorts | Pre-<br>conditioning<br>(FLU-CY; Days<br>-6, -5, -4, -3) | Total CD19/CD22<br>CAR-Positive T<br>Cells (Day 0) | Regimen A:<br>Consolidation<br>(pembrolizumab; Days<br>14, 35, 56) | Regimen B:<br>Pre-conditioning<br>(pembrolizumab; Day -<br>1) |
|---|---|---|---|---|---|
| Dose<br>Level 1 | Cohort 1 | Yes | 50 x 10 <sup>6</sup> | None in first 3 patients,<br>then Yes | |
| Dose<br>Level 2 | Cohort 2A | Yes | 150 x 10 <sup>6</sup> | Yes | |
| Dose | Cohort 3A | Yes | 450 x 10 <sup>6</sup> | Yes | |
| Level 3 | Cohort 3B | Yes | 450 x 10 <sup>6</sup> | | Yes |



Final 1.0/ 21-Dec-2023

| Dose<br>Levels | Treatment<br>Cohorts | Pre-<br>conditioning<br>(FLU-CY; Days<br>-6, -5, -4, -3) | Total CD19/CD22<br>CAR-Positive T<br>Cells (Day 0) | Regimen A:<br>Consolidation<br>(pembrolizumab; Days<br>14, 35, 56) | Regimen B:<br>Pre-conditioning<br>(pembrolizumab; Day -<br>1) |
|---|---|---|---|---|---|
| Dose | Cohort 4A | Yes | 900 x 10 <sup>6</sup> | Yes | |
| Level 4 | Cohort 4B | Yes | 900 x 10 <sup>6</sup> | | Yes |
| RP2D | RP2D or<br>Dose Range<br>Cohort | Yes | 150 to 450 × 10 <sup>6</sup> | | Yes |
| CAR=Chir | | eceptor: FLU-CY= | <br>Fludarabine and Cvclo | <br>phosphamide; RP2D=recomi | mended Phase II dose. |

A few important aspects considered for the planned dose decision are listed below:

- In dose level 1, the first three patients treated at 50 × 10<sup>6</sup> CD19/CD22 CAR-positive T cells will not receive consolidation with pembrolizumab.
- Consolidation therapy with pembrolizumab (except dose on Day -1) will be administered
  only after any CRS has resolved to ≤ Grade 1 or NT has resolved. Based on emerging data,
  either one or both pembrolizumab dosing regimens will be opened in Dose Level 4 (Cohorts
  4A and 4B).
- On occasion, AUTO3 production may fail to generate sufficient cells for the current dose level. In this case, the patient can be treated on study but at a lower dose, however if production fails to generate ≥15 × 10<sup>6</sup> (approx. 0.2 × 10<sup>6</sup>/kg) CD19/CD22 CAR-positive T cells, near the lowest known active dose of CD19 CAR-positive T cells (1.46 × 10<sup>5</sup> T cells/kg, approximately total dose of 10 × 10<sup>6</sup> T cells), then the patient will not be treated on the study. Only patients treated at planned dose level will be evaluable for dose escalation decision making and primary efficacy analysis (± 20% window). Additional patients will be treated to meet the minimum number needed to make the dose escalation decision.
- If emerging data suggest that escalation is appropriate to an intermediate dose, which is a lower than the planned dose, then it can be undertaken with Regimen A or B. Total number of patients of Phase I may also be increased if necessary.
- If emerging safety and efficacy data suggest further dose escalation is warranted, any doses higher than  $900 \times 10^6$  CD19/CD22 CAR T cells will not be undertaken without a substantial



Final 1.0/ 21-Dec-2023

protocol amendment.

<u>Note:</u> The dose determination is based solely upon the genetically modified cells (i.e. CD19/CD22 CAR-positive T cells). A patient may be eligible for a planned dose level if the dose is within ±20% of the prescribed CD19/CD22 CAR-positive T cells dose.

<u>Phase I expansion cohort:</u> In this cohort, the safety and tolerability of AUTO3 at the RP2D or dose range will be assessed in an outpatient/ambulatory care setting following declaration of RP2D or dose range in the dose escalation part. Approximately 20 patients will be treated. There will be no inter-patient dosing interval.

Patients enrolled in this cohort will be monitored for at least 10 days in an outpatient/ambulatory care setting, or until all AUTO3-non-haematological related toxicities have returned to Grade ≤1 or baseline, or longer as clinically necessary. During the 10 days following AUTO3 infusion, the patients are monitored at a minimum every 2 to 3 days (in the UK, at least once a day evaluation by a physician or qualified designee). In addition, it is recommended for the patient to have a daily verbal communication with qualified nurse/medical personnel (phone call). Patients will also need adequate caregiver support (in line with institutional outpatient transplant guidelines). Patients enrolled or treated in this cohort can be admitted to the inpatient setting as necessary for the management of AEs or toxicity at any time. Patients can also be admitted based on Investigator discretion should they consider it inappropriate to treat or monitor an already enrolled patient in an outpatient/ambulatory setting. Physicians may also admit patients for social reasons. In all cases the reason for admission should be documented.

<u>Phase II dose expansion:</u> Once the RP2D(s) or dose range is/are determined, the Phase II dose expansion part of the study will open with two cohorts. This part will treat approximately up to 101 patients on the RP2D(s). Cohort 1 will comprise approximately 81 patients on the RP2D with DLBCL subsets and transformed FL, Cohort 2 will comprise approximately 20 patients with PMBCL and DLBCL transformed from other indolent histologies. Patients treated at a dose lower than the RP2D(s) will not be evaluable for primary efficacy endpoint analysis but will be evaluable for secondary efficacy endpoints and safety analysis. Once Phase II starts, patients can be dosed simultaneously at the declared RP2D dose(s) without inter-patient intervals.

# 5.3 RANDOMISATION AND BLINDING

Randomisation will not be used in this study. As this is an open-label study, blinding procedures are not applicable.



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

#### 5.4 SAMPLE SIZE JUSTIFICATION

Approximately 171 patients in total are expected to be enrolled (consented) into both the dose escalation and expansion parts of the study, and approximately 151 patients in total are anticipated to be treated with AUTO3 therapy.

Phase I (Escalation): Up to 30 patients treated (3 to 6 patients per dose cohort, with the
exception of dose level cohort 1 one which may include up to 12 patients [up to 6
patients without anti-PD-1 treatment, and 6 patients with anti-PD-1 treatment]),
following a rolling 6 design (Skolnik et al. 2008).

An additional 12 patients may be added to RP2D dose /dose range.

 Phase I Expansion Cohort: Approximately 20 patients will be treated in an outpatient/ambulatory care setting.

At the end of Phase I (Escalation), assuming at least 12 patients are treated, the study will terminate if the upper limit of the 2-sided 95% confidence interval in response rate is less than 30%. This is equivalent to observing 0 response in 12 patients. The study will proceed to Phase II if the upper limit of the 2-sided 95% confidence interval in response rate exceeds 30%.

Phase II: In cohort 1, up to 81 evaluable patients will be analysed, using Simon's 2-stage optimal design. This will include 81 patients with DLBCL (and its defined subsets), and those with transformed FL. Additionally, 20 patients with primary mediastinal large B cell lymphoma and those with lymphoma transformed from other indolent histologies will be enrolled in Cohort 2.

Simon's two-stage design trial will be used (Simon 1989) in the Phase II Cohort 1 only. The null hypothesis that the true response rate is 30% will be tested against a 1-sided alternative. In the first stage, 27 evaluable patients will be accrued. If there are 9 or fewer responses in these 27 patients, the study will be stopped.

Otherwise, 54 additional evaluable patients will be accrued for a total of 81 in Cohort 1. The null hypothesis will be rejected if 31 or more responses are observed in 81 patients. This design yields a type I error rate of 5% and 80% power when the true response rate is 45%.



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

# 6 Statistical Considerations

6.1 TERMINATION OF THE STUDY AFTER END OF PHASE I

# <u>Important Note – Early Study Termination:</u>

Sponsor informed Cmed team on 03Nov2021 that it was decided not to progress AUTO3 DB1 study into the Phase II part of the study.

Over a period of 4 years (2017-2021), a total of 73 patients were enrolled and 52 patients received AUTO3 in the Phase I part of the study. After reviewing the data and taking into consideration the available treatment landscape in r/r DLBCL, Autolus has decided not to progress AUTO3-DB1 into the Phase II part of study. Therefore, the study will be terminated after the completion of Phase I and not progress to Phase II.

The SAP documents were initially drafted including details for Phase I/Phase II and Interim Analyses for Phase I/Phase II. The study will now focus the analysis only on Sponsor's requirements for end of the study for Phase I only.

6.2 SOFTWARE

The SAS Viya 3.5 (or higher), will be used for all analysis, unless otherwise specified.

6.3 MISSING DATA HANDLING

No other imputation for missing data will be carried out other than to complete partial dates using standard imputation techniques as described below.

For the time to event variables censoring rules will apply as defined in <u>section 8.12</u>, so there should be no missing data.

# 6.4 PARTIAL DATE IMPUTATION

The following rules should be used when modifying partial or missing dates for reporting purposes such as defining on treatment flags.



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

A permanent new date variable should be created if there is a requirement to be used in determining flags, sort orders and other derived variables needed for a table, listing or figure. Imputed date variable names will be defined in the derived dataset specifications.

Original (raw) date variables must not be overwritten. Imputed dates will not be displayed in the listings.

Database does not allow adverse events to have any partial dates.

General rules

**Prior/Concomitant Medications or Prior Cancer Therapies / Bridging Therapies** 

Prior/concomitant medications and prior cancer therapies/bridging therapies are considered to have started at the earliest possible date and end at the latest possible date.

In case of partial start dates with missing day:

 Any partial start date in the same month as the AUTO3 infusion would be imputed at the date of the AUTO3 infusion.

Any partial start date in the month before AUTO3 infusion and in the same month as
pre-conditioning treatment would be imputed at the date of earliest pre-conditioning
treatment date during that month.

Any partial CM start date would be imputed at the first day of the month, regardless
of if during the same month as pre-conditioning or AUTO3 infusion.

 Any partial start date after the month of AUTO3 infusion would be imputed at the first day of the month.

 Any partial start date before the month of first AUTO3 infusion and before the month of first pre-conditioning treatment would be imputed at the last day of the month.

In case of partial start dates with missing day and missing month:

 Any partial start date during the year of AUTO3 infusion would be imputed at the date of the AUTO3 infusion.

 Any partial start date before the year of first AUTO3 infusion and during the year of preconditioning treatment would be imputed at the date of earliest pre-conditioning



Final 1.0/21-Dec-2023

treatment date during that year.

- For any concomitant medication or further treatments starting before or during the year of AUTO3 infusion, the start date would be imputed at 01 January of that year.
- For any concomitant medication or further treatments starting after the year of first
   AUTO3 infusion, the start date would be imputed at 01 January of that year.
- For any concomitant medication or further treatments started before the year of first AUTO3 infusion and before the year of first pre-conditioning treatment, the start date would be imputed as the 31 December of that year.

In case of partial end dates with missing day:

 Partial end dates would be imputed at the last day of the month or at the date of study discontinuation, whichever occurs first.

In case of partial end dates with missing day and month:

 Partial end dates would be imputed at the last day of December (i.e. 31st December) or at the date of study discontinuation, whichever occurs first.

Some examples are given below (YYYY-MM-DD).

In most cases, start dates are imputed as first day of the month or first of January.

| Data Type | Start Date | Imputed<br>Start Date | First pre-<br>condition<br>treatment<br>date | Last pre-<br>condition<br>treatment<br>date | First AUTO3<br>infusion date | End Date | Imputed End<br>Date |
|---|---|---|---|---|---|---|---|
| Prior/Concomitant<br>Meds/Further<br>treatments | 2017-02 | 2017-02-<br>01 | 2016-12-11 | 2016-12-13 | 2016-12-17 | 2017-02 | 2017-02-29 |
| Prior/Concomitant<br>Meds/Further<br>treatments | 2017-02 | 2017-02-<br>01 | 2017-01-27 | 2017-01-29 | 2017-02-03 | 2017-02 | 2017-02-29 |
| Prior/Concomitant<br>Meds/Further<br>treatments | 2017-02 | 2017-02-<br>11 | 2017-02-11 | 2017-02-13 | 2017-02-18 | 2017-02 | 2017-02-29 |
| Prior/Concomitant<br>Meds/Further<br>treatments | 2017-02 | 2017-02-<br>03 | 2017-01-27 | 2017-01-29 | 2017-02-03 | 2017-03 | 2017-03-31 |



Sponsor: Autolus
Protocol: AUTO3-DB1
Statistical Analysis Plan:
Final 1.0/ 21-Dec-2023

| Prior/Concomitant<br>Meds/Further<br>treatments | 2017 | 2017-01-<br>27 | 2017-01-27 | 2017-01-29 | 2017-02-03 | 2017 | 2017-03-16 £ |
|---|---|---|---|---|---|---|---|
| Prior/Concomitant<br>Meds/Further<br>treatments | 2017-03 | 2017-03-<br>01 | 2017-01-27 | 2017-01-29 | 2017-02-03 | 2017-03 | 2017-03-31 |
| Prior/Concomitant<br>Meds/Further<br>treatments | 2017-01 | 2017-01-<br>27 | 2017-01-27 | 2017-01-29 | 2017-02-03 | | 2017-03-01 * |
| Prior/Concomitant<br>Meds/Further<br>treatments | 2017-01 | 2017-01-<br>31 | 2017-02-27 | 2017-02-29 | 2017-03-03 | 2017-01 | 2017-01-31 |

£ patient discontinued on 2017-03-16; \* patient discontinued on 2017-03-01.

# **Date of Diagnosis**

Partial dates for initial diagnosis will be imputed as the 15th of the month if the month is present, or the 1st of July if only the year is present.

# **Response Assessment**

Partial dates are not expected for response assessment data. However, should partial dates be present on treatment disease assessments:

- First of the month or the date of AUTO3 infusion (whichever is later) if the day part is missing, but month and year parts are present.
- First of January or the date of AUTO3 infusion (whichever is later) if the day and month parts are missing, but year part is present.

#### Death

Partial dates are not expected for deaths. However, in case of partial date for death, the date would be imputed as:

- The day after the last visit/assessment date when the patient was known alive, if the death date is completely missing, or if the month and year parts are the same as the month and year parts of the last visit/assessment date.
- First of the month if the day part is missing, but month and year parts are present.
- First of January if the day and month parts are missing, but year is present.



Final 1.0/ 21-Dec-2023

# 6.5 VISIT WINDOWING

Planned assessments will not be re-assigned to any planned visits using statistical programming based on assessment date. All the data will be analysed according to the planned visit as collected in the eCRF.

# 6.6 BASELINE

Baseline is defined as the last non-missing value/result where assessment date is less than or equal to the date of first pre-conditioning treatment, unless otherwise specified for individual assessments. Baseline will be determined based on all assessments, including additional assessments.

Change from baseline is defined as the difference between the post-baseline assessment value and the baseline value.

# 6.7 REPORTING GUIDELINES

The following guidelines will be followed:

- Page Orientation: Landscape.
- **Post-text TFLs**: will be generated in .rtf using ods rtf within SAS.
- For final delivery TFLs will be provided in combine files.
- No in-text outputs are planned.
- Font: TFLs will use Courier New font with minimum of 8 point font size.
- Margins: Left: 2 cm, Right: 2 cm, Top: 2 cm, Bottom 2 cm on letter paper.
- Columns header will be left aligned.
- Treatment labels for Phase I will be the following and displayed in the following order, unless otherwise stated:
  - 50x10^6 (No Pem)
  - 50x10^6 (D14 Pem)
  - 150-450x10^6 (D14 Pem)



Sponsor: Autolus
Protocol: AUTO3-DB1
Statistical Analysis Plan:
Final 1.0/ 21-Dec-2023

- o 150-450x10^6 (D-1 Pem) Inpatient
- o 150-450x10^6 (D-1 Pem) Outpatient
- All summaries and analyses will be presented by the actual dose, unless otherwise stated.
- Visit labels: the visit labels displayed in <u>Table 2</u> will be used as required.

**Table 2: Visit Labels** 

| Study Stage | CRF Visit | Tables, Figures and Listings<br>Label |
|---|---|---|
| | Screening 1: Day -84 to -35 | Screening 1 |
| Screening and<br>Leukapheresis | Leukapheresis: Day -84 to -35 | Leukapheresis |
| Leukapheresis | Screening 2: Day -35 to -6* | Screening 2 |
| | Pre-conditioning Day -5 | PRE-COND Day -5 |
| Pre-conditioning | Pre-conditioning Day -4 | PRE-COND Day -4 |
| | Pre-conditioning Day -3 | PRE-COND Day -3 |
| | Day -1 to Day 0** | Day -1 to 0 |
| | Day 1 | Day 1 |
| | Day 3 | Day 3 |
| | Day 4 | Day 4 |
| | Day 5 | Day 5 |
| | Day 7 | Day 7 |
| AUTO 3 Treatment & | Day 9 | Day 9 |
| Anti-PD-1 Consolidation | Day 10 | Day 10 |
| phase# | Day 12 | Day 12 |
| | Day 14 | Day 14 |
| | Day 16 | Day 16 |
| | Day 18 | Day 18 |
| | Day 20 | Day 20 |
| | Day 28 | Day 28 |
| | Day 35 | Day 35 |



Final 1.0/ 21-Dec-2023

| Study Stage | CRF Visit | Tables, Figures and Listings<br>Label |
|---|---|---|
| | Day 41 | Day 41 |
| | Day 56 | Day 56 |
| Re-Treatment Pre-<br>conditioning phase | Re-Treatment Pre-conditioning Day -5 | Re-TRT PRE-COND Day -5 |
| | Re-Treatment Pre-conditioning Day -4 | Re-TRT PRE-COND Day -4 |
| | Re-Treatment Pre-conditioning Day -3 | Re-TRT PRE-COND Day -3 |
| Re-Treatment AUTO 3<br>Treatment & Anti-PD-1<br>Consolidation phase *** | Re-Treatment Day -1 to Day 0 | TRT Day -1 to Day 0 |
| | Re-Treatment Day 1 | Re-TRT Day 1 |
| | Re-Treatment: Day 4 | Re-TRT: Day 4 |
| | Re-Treatment Day 56 | Re-TRT Day 56 |
| Follow-up phase<br>Efficacy & Safety Follow-<br>up# | Follow-up: Month 2 | FU (M2) |
| | Follow Up: Month 3 | FU (M3) |
| | Follow Up: Month 4 | FU (M4) |
| | Follow Up: Month 5 | FU (M5) |
| | Follow Up: Month 6 | FU (M6) |
| | Follow Up: Month 9 | FU (M9) |
| | Follow Up: Month 12 | FU (M12) |
| | Follow Up: Month 15 | FU (M15) |
| | Follow Up: Month 18 | FU (M18) |
| | Follow Up: Month 24 | FU (M24) |
| | Efficacy/Safety Month 30 | FU (M30) |
| | Efficacy/Safety Month 36 | FU (M36) |
| | Efficacy/Safety Month 42 | FU (M42) |
| | Efficacy/Safety Month 48 | FU (M48) |
| | Efficacy/Safety - End of Study | End of Study |

<sup>\*</sup>Pre-conditioning assessment Day-6 will be covered under Screening 2: Day -35 to -6.

Note: Visits from 'Safety and Survival Follow-up' phase are captured as unscheduled visits.

<sup>\*\*</sup> Pre-conditioning assessment Day-1 will be covered under Day -1 to Day 0.

<sup>\*\*\*</sup>Days corresponding to the visits during the Re-Treatment phase are same as the weeks corresponding to the visits during the Treatment phase.

<sup>#</sup> Under 'AUTO 3 Treatment & Anti-PD-1 Consolidation' and 'Follow-up' phases all visits will be reported as per database, depending on which protocol version was followed when the assessment was performed.



Final 1.0/ 21-Dec-2023

- Unscheduled visit / repeat assessments /disease assessment visits: Data obtained at
  unscheduled or repeat assessments will be included in time to event analyses, baseline
  determination and anti-tumor effect. All other data from unscheduled or repeat
  assessment will not be included in summaries but only be presented in data listings, if
  not otherwise specified.
- Data collected during <u>re-treatment</u> will only be listed, if not otherwise specified.
- **N:** The number of patients in the specified population and cohort.
- **Treatment presentation:** Generally, data will be summarized separately for all data available, unless otherwise specified. The summaries will be presented as follows:
  - 50x10^6 (No Pem)
  - 50x10^6 (D14 Pem)
  - o 150-450x10^6 (D14 Pem)
  - o 150-450x10^6 (D-1 Pem) Inpatient
  - 150-450x10^6 (D-1 Pem) Outpatient
  - Overall
- Continuous data will be summarized using number of patients (n), mean, standard deviation (SD), median, minimum value, maximum value and number of missing data (if there are any). For time to event summaries, median, quartiles (Q1 and Q3) and corresponding 95% confidence interval (CI) for the median and quartiles will be presented.
- **Categorical data** will be summarized using n and percentage based on number of non-missing data.
  - All categories will be presented, even if no patients are counted in a particular category.
  - In case 1 or more patients have missing data for the summary, the number of missing data will be presented as a separate category, labelled accordingly as 'Missing', if not otherwise stated.
  - o Counts of zero in any category will be presented without percentage.
  - All summaries percentages will be calculated using the number of patients with an assessment, unless otherwise stated.
  - For AEs, medical history, prior and concomitant medications the counts are based on single counts of patients with multiple events/treatments under same category, while the percentages are calculated using N.



Final 1.0/ 21-Dec-2023

# Precision of summary statistics:

- Integer Sample size (n, N) and number of missing data (if displayed);
- One additional decimal place than reported/collected mean, median, other percentile, confidence interval;
- Two additional decimal places than reported/collected standard deviation;
- Same number of decimal places as reported/collected minimum, maximum;
- Percentages one decimal place.
- Study day, as per visit schedule is calculated with reference to first AUTO3 infusion date as Day 0 for consistency with the protocol. This study day is not used for TFLs.
- Study day, for inclusion in CDISC compliant datasets and TFLs will be calculated with reference to first AUTO3 infusion date as Day 1. It will be included in CDISC compliant datasets only and will be displayed in TFLs. This will be calculated as (assessment date date of first AUTO3 infusion) +1 if it's on or after first date of AUTO3 infusion, or (assessment date date of first AUTO3 infusion) if it is prior to AUTO3 infusion.
- **DLT period:** 28 days after the infusion of AUTO3 or at least 14 days after the first dose of pembrolizumab, if administration of first pembrolizumab dose is delayed beyond Day 14.
- Data will be presented in listings by cohort. The order will be subject ID, visit, assessment date/time and assessment type/parameters (in order collected on e-CRF, unless otherwise specified). In case of clinical laboratory results, the listings will be presented in order cohort/group, subject ID, parameter, assessment date/time, visit.
- Dates will be presented in format YYYY-MM-DD.
- Version 5.0 of the NCI-CTC grading criteria (CTCAE v5) will be used for relevant tables.
- Latest version of the Medical Dictionary for Regulatory Activities (MedDRA) will be used for relevant tables. The version will be documented in the footnote of the corresponding TFLs.
- Latest version of the WHO-DD/DDE dictionary will be used for prior and concomitant medication coding. The version will be documented in the footnote of the corresponding TFLs.
- File naming: Each TFL output file will be named with a t, I or f to denote the output type and then according to its table numbering.



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

# 7 Analysis Sets

7.1 ANALYSIS SETS

#### Screened set

The screened set will consist of all patients who have signed informed consent and were screened in the study.

# Safety set

All patients who received at least 1 dose of AUTO3 therapy will be included in the safety set.

#### Infused set

All patients who received at least 1 dose of AUTO3 therapy will be included in the infused set. This is the same as the safety set.

# **Evaluable set**

All patients who received at least 1 dose of AUTO3 therapy and had FDG PET scan positive disease prior to pre-conditioning.

# 7.2 PROTOCOL DEVIATIONS

The full list of types of protocol deviations (PDvs) and their relation to the analysis sets, along with the method of identification of each protocol deviation, are detailed in the protocol deviation criteria form which is separate to this SAP. This will be used as a basis for identifying patients with protocol deviations throughout the study.

Protocol deviations noted during the trial will be tracked throughout the study by Autolus. The PDvs will be read into SAS® prior to reporting.

Prior to database lock, PDvs will be reviewed and agreement of the final analysis populations made.

Important protocol deviations will be summarized by deviation category on the Screened set. A listing of all confirmed reported protocol deviations (with both Important PD = Yes or No) by patient will also be provided along with the deviation category, verbatim term and deviation



Final 1.0/ 21-Dec-2023

date.

# 8 Methods of Analyses and Presentations

# 8.1 PATIENT DISPOSITION

The patient disposition summaries will be presented on overall group using the Screened set.

The summary of patient disposition will be showing the number and percentages of patients belonging to the following categories:

- Discontinued before leukapheresis (and reasons)
- Leukapheresed
  - o Discontinuation prior AUTO3 infusion (and reasons)
  - AUTO3 infused

Patients in analysis populations will be summarized.

Information on analysis populations, study completion and discontinuation will also be displayed in patient listings.

# 8.2 DEMOGRAPHIC AND BASELINE CHARACTERISTICS

The following demographic and baseline characteristics will be summarized on the Infused set:

- Age;
- Age group (<65 years, ≥65 years);</li>
- Gender;
- Race;
- Ethnicity;
- Weight;
- ECOG performance at study entry.



**Sponsor**: Autolus **Protocol**: AUTO3-DB1

Final 1.0/ 21-Dec-2023

**Statistical Analysis Plan:** 

Also, the following lymphoma disease characteristics will be summarized, on the Infused set:

- Current lymphoma subtype:
  - Current stage of lymphoma;
  - Current lymphoma subtype;
- Relapsed and/or refractory disease.
- International Prognostic Index (IPI).
- Extranodal disease at baseline.
- Molecular Subtype [Note: This will be available for the patients consented to the study under Protocol amendment 7 (onward)].
- Sum of product of perpendicular (SPD) diameters prior to pre-conditioning.
- Lactate dehydrogenase (LDH) prior to pre-conditioning.

Listings of all demographic and baseline characteristics data will be produced.

# 8.3 PRIOR LYMPHOMA THERAPIES

Listings of all prior lymphoma therapies and medications along with best response result will be produced. A separate listing with prior lymphoma radiotherapy will be presented. In addition, a listing containing prior stem cell transplant (SCT) details will be also presented.

The following summaries will be presented on the Infused set:

- Lines of therapies (summarized through summary statistics and number and percentages of patients with 1, 2, 3, 4, >=5 lines)
- Number and percentages of patients with prior SCT.

# 8.4 MEDICAL HISTORY

Medical histories and concomitant diseases will be coded using MedDRA. Summaries of patient medical histories and concomitant diseases will be produced on the Infused set, by system organ class and MedDRA preferred term by cohort and overall.

Listing of medical history will be produced. Also, a separate listing presenting surgical and medical procedures will be provided.



Final 1.0/ 21-Dec-2023

# **8.5 PRIOR AND CONCOMITANT MEDICATIONS**

Medications other than the study treatment (including leukapheresis related medications, preconditioning related medications and AUTO3 related medications) will be coded using the WHO-DD/DDE dictionary. Medications will be defined as follows:

- Prior Medication: Any medication whose medication start date is before the first AUTO3 infusion date.
- Concomitant Medication: Any medication whose medication start or end date is either the same as or after the first AUTO3 infusion date.

Any medication with a missing medication end date will be assumed to be concomitant medication. Also, ongoing medications are considered as concomitant medications. A medication can be both a prior and a concomitant medication.

Summaries of prior medications and concomitant medications will be produced by ATC class and preferred term on the Infused set.

Medications defined as both prior and concomitant will appear in both tables.

In addition, a listing of prior and concomitant medications will be presented.

# 8.6 BRIDGING THERAPIES AND NEW ANTI-CANCER THERAPIES

Bridging therapies (therapies between informed consent up to AUTO3 dosing) and new anticancer treatment (anti-cancer medications or new anti-cancer radiotherapy) post AUTO3 infusion will be presented in separate listings.

Bridging therapies will be summarized by ATC class and preferred term on the Infused set.

# 8.7 IMMUNOGLOBULIN THERAPIES

Intravenous immunoglobulin therapy (IVIG) can also be administered to the patients, if needed.

Immunoglobulin administration details will be presented in a listing.

#### 8.8 LEUKAPHERESIS

A listing of leukapheresis details will be presented. Leukapheresis related medications will be presented and summarized with the prior and concomitant medications.



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

# 8.9 LYMPHOMA B-SYMPTOMS

The lymphoma B-symptoms at baseline (Screening) and at post-treatment visits will be listed on the Screened set.

### 8.10 STUDY TREATMENT

# Pre-Conditioning: Fludarabine and Cyclophosphamide

The number and percentage of patients who received at least one dose of the pre-conditioning regimen will be summarized by medication received in the Safety set. Duration of exposure (days) will also be summarized.

A listing of pre-conditioning treatment administration with Fludarabine and Cyclophosphamide will be presented.

# **Study treatment: AUTO3**

Days from leukapheresis to first AUTO3 infusion will be calculated as [(Date of first AUTO3 treatment – Date of last leukapheresis) + 1] and summarized.

For AUTO3 infusion exposure summary statistics will be presented for the following:

- Number of patients treated with AUTO3;
- Number of patients re-treated with AUTO3;
- Number of cells administered to the patient.

Details of AUTO3 infusion administration and treatment exposure, including re-treatment details will be listed.

# **Consolidation Treatment: Pembrolizumab**

A listing of anti-PD-1 consolidation treatment administration with pembrolizumab (Regimen A and Regimen B) will be presented.

# 8.11 FOLLOW-UP TIMES

Follow-up time will be calculated for each patient using the following formula:



Protocol: AUTO3-DB1
Statistical Analysis Plan:

Final 1.0/ 21-Dec-2023

Follow-up time (months) = [(Date of last follow-up visit when patient was known alive (or date of death (if applicable)) – Date of first AUTO3 treatment) + 1]/ 30.4375 days

Time from first AUTO3 treatment to data extraction or LPLV (as applicable) and time from leukapheresis to first AUTO3 treatment will be presented.

Follow-up times will be summarized on the Infused set.

# 8.12 EFFICACY DATA ENDPOINTS AND ANALYSES

Disease evaluation will be performed to assess disease status at end of DLT period (Day 28), Month 3, Month 6, Month 9, Month 12, and yearly until end of study. Note, the baseline assessment should be performed within 35 days of starting pre-conditioning (approximately 40 days before receiving AUTO3). Patients receiving bridging therapy should have the baseline disease assessment after the bridging therapy is completed and prior to starting pre-conditioning. All post-baseline response assessments will be considered for the analyses (unless otherwise stated).

In Phase I disease response will be assessed by investigators.

All time to event efficacy endpoints defined in <u>section 8.12.2</u> will be calculated in days and converted to months considering the following conversion: 1 month = 30.4375 days.

Efficacy data will be summarized on the Infused set, unless otherwise specified.

A listing will be provided detailing the disease status, response and progression for each patient at each visit. Disease assessment will be listed. Also, all efficacy endpoints defined as below will be listed.

# 8.12.1 Primary Efficacy Endpoint and Analyses

# 8.12.1.1 Anti-tumour effect of AUTO3

Primary efficacy analysis is based on whether a patients achieved an objective response post AUTO3 infusion. An objective response is defined as a complete response (CR) or partial response (PR) post AUTO3 infusion.

The best overall response (BOR) is the first best response (CR>PR>SD>PD>NE)\* recorded from



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

the first post-baseline (post-AUTO3 infusion) assessment until end of study, as assessed by the investigators.

\*CR=Complete response, PR=Partial response, SD=Stable disease, PD=Progressive disease, NE=Not evaluable.

Patients who do not have any post-baseline assessments will be classified as having BOR of Not evaluable (NE).

Best overall response post-AUTO3 infusion will be summarized by presenting the number and percentages of patients with each type of best overall response assessed from all assessments post-AUTO3 infusion. The overall response rate will be presented. This is defined as the numbers of responders (CR and PR) out of the number of patients treated with AUTO3.

In summary, the following counts will be presented:

- Number of responders [objective response]: CR+PR.
- Number of patients by each response: CR, PR, SD, PD, NE

The percentage calculation will be based on N.

BOR will be presented on the Evaluable set.

# 8.12.2 Secondary Efficacy Endpoints and Analyses

# 8.12.2.1 Duration of response

Duration of response (DOR) is defined as the time from the first observed CR or PR [from the first post-baseline response assessment] until the date of first progressive disease or death due to underlying cancer (primary reason for death=progressive disease), whichever occurs first. Only responders (patients with BOR of CR or PR) will be included in the analysis of duration of response.

Patients with death not due to underling cancer (primary reason for death=AE or Other or Unknown) or who received new anti-cancer therapy other than SCT or discontinued from the study for other reason than PD or who are lost to follow-up or reach the time point of analysis without a known record of progression or death will have the duration of response censored at the date of last adequate disease assessment for response.

Patients who received a new SCT will be censored at the start date of this new date of SCT, if the

Template Author:


BMSOP111/F2

Version 5.0 25Jun2020



**Sponsor**: Autolus **Protocol**: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

patients have not already had disease progression recorded.

Estimates of the survival function for DOR (median [95% CI], Q1 [95% CI] and Q3 [95% CI]) will be obtained using the Kaplan-Meier method. The CI for the median will be calculated using the Brookmeyer and Crowley method. The survival function and associated 95% CI at relevant timepoints will also be presented. The CI will be obtained using the Kaplan-Meier method and a log-log transformation for CI (SAS PROC LIFETEST CONFTYPE=LOGLOG). The final choice of the time points presented in the life table might be updated dependent upon the data at the time of the analysis. DOR will also be presented graphically. DOR will be listed.

# 8.12.2.2 Progression-Free Survival

The progression-free survival (PFS) is defined as the time from first AUTO3 treatment until the first progression of disease or death from any cause, whichever occurs first.

Patients who reach the time point of analysis without a known record of progression will have the PFS censored at the date of last adequate disease assessment.

Patients who received a new SCT will be censored at the start date of this new SCT.

Patients who received a new anti-cancer therapy or discontinued from the study for other reason than PD and who are lost to follow-up will be censored at the date of last adequate disease assessment.

For patients with no post-baseline disease assessments a censored PFS at day 1 will be considered.

Estimates for the survival function for PFS will be summarized and presented graphically, similarly as the DOR. Also, PFS will be listed.

Swimmer plot of PFS will be presented.



Final 1.0/ 21-Dec-2023

#### 8.12.2.3 Overall Survival

Overall survival (OS) is defined as the time from the date of first AUTO3 treatment up to the date of death, regardless of cause of death.

Patients alive at the time of the analysis will have the OS censored at the date of last assessment when the patient was known alive.

Date of last assessment patient is known alive will be determined based on vital sign, laboratory (hematology and biochemistry), immunoglobulin, lesions (target, non-target, new), blood samples (cytokines, PK, PD, biomarker), adverse events, concomitant medications and ECOG assessments. For patients in the follow-up period, date of last assessment is based also on date of last contact when patient was known alive (e.g. last contact could be telephone contact).

For patients with no post-baseline assessments a censored OS at day 1 will be considered.

Estimates for the survival function for OS will be summarized and presented graphically similarly as the DOR. OS will be listed.

8.12.2.4 Biomarker expression of PD-L1, CD19 and CD22

CD19 and/or CD22 relapse analysis will be covered in PK/PD SAP, outside of this SAP.

# 8.12.3 Exploratory Efficacy Endpoints and Analyses

8.12.3.1 Time course and magnitude of cytokine release

Individual spaghetti plots for the cytokine levels will be presented over time by treatment groups for each patient for each parameter. Boxplot of peak cytokine level per patient will be also presented per treatment group.

# 8.12.4 Additional Efficacy and Biomarker Assessments

The following measurements are essential in establishing the clinical efficacy of AUTO3 and associated response on which the primary and secondary efficacy endpoints are based, as described in section 8.12.1 and section 8.12.2.

The following assessments will be listed:


Final 1.0/ 21-Dec-2023

- Immunoglobulin results: IgG, IgA, IgM;
- •
- Flow cytometry for B cells as assessed at specific timepoints to characterize the duration of B cell aplasia;
- RCR testing and insertional mutagenesis.

#### 8.12.5 Subgroup Analysis

Not applicable.

#### 8.13 PHARMACODYNAMIC AND PHARMACOKINETIC ENDPOINTS AND ANALYSES

All pharmacokinetics and pharmacodynamic analysis will be performed by Sponsor.

## 8.14 QUALITY OF LIFE OR PHARMACOECONOMIC ENDPOINTS AND ANALYSES

Not applicable.

#### 8.15 SAFETY DATA ENDPOINTS AND ANALYSES

#### 8.15.1 Adverse Events (AEs)

Adverse events will be coded using the MedDRA coding system. The version of the dictionary will be provided in the adverse events TFLs footnotes.

#### AUTO3 TEAE is defined as any AE with onset during the post AUTO3 infusion period.

AEs that are considered related to Cyclophosphamide, Fludarabine, pembrolizumab and/or AUTO3 treatment (possibly, probably, or definitely related) will be collected accordingly on the eCRF.

Any AE that is present at baseline but worsens in intensity after the first dose of study treatment should be entered into the eCRF as a different AE record with the differing grade recorded.

The number and percentage of patients will be summarized by System Organ Class (SOC) and Preferred Term (PT) by all grades (1-5) and grade >=3. Patients will be counted only once within each SOC and PT by dose level. SOCs will be sorted by alphabetical order of frequency for each

Template Author: Andra Rusu  BMSOP111/F2

Version 5.0 25Jun2020



Final 1.0/ 21-Dec-2023

group, PTs will be sorted by descending order of frequency for each group within each SOC. The following summaries will be presented:

- AUTO3-TEAEs, within 75 days (i.e. occurring on study days 1 through 75) and anytime post infusion
- AUTO3-TEAEs, related to AUTO3 treatment, within 75 days and anytime post infusion
- AUTO3-TEAEs, specific AEs (i.e. Neutropenia or Neutrophil count decreased, Thrombocytopenia or Platelet count decreased, Anemia or Hemoglobin count decreased, Infections (including all SOC Infections and infestations)) within 30 days, within 75 days and anytime post infusion
- CRS
- Neurotoxicity [(Protocol amendments 1-7)]
- Serious AUTO3-TEAEs, within 75 days, and anytime post infusion
- Non-serious AUTO3-TEAEs, within 75 days and anytime post infusion
- Fatal TEAEs (i.e. grade 5 toxicity TEAEs), within 30 days (i.e. occurring on study days 1 through 30) and anytime post infusion

In addition, the number and percentage of patients will be summarized by Preferred Term (PT) by all grades (1-5) and by grade >=3. Patients will be counted only once within each PT by dose level. PTs will be sorted by descending order of frequency for the overall group. The following summaries will be presented within 75 days and any time post infusion:

- AUTO3 TEAEs
- AUTO3-TEAEs, related to AUTO3 treatment
- Serious AUTO3-TEAEs
- Non-serious AUTO3-TEAEs

All summaries will be presented on the Safety set.

All information on AEs will be listed. A separate listing of SAEs will be provided.

#### 8.15.1.1 CRS AEs

The number and percentage of patients with CRS events along with the maximum CRS grade will be summarized.

Time to onset of the first CRS event post AUTO3 infusion, defined as the time from first AUTO3 infusion until the date of first CRS event, will be presented.

Template Author:
Version 5.0 25Jun2020



Sponsor: Autolus
Protocol: AUTO3-DB1
Statistical Analysis Plan:
Final 1.0/ 21-Dec-2023

Similarly, time to onset for the first Grade 3 or above CRS will be presented.

Duration of CRS events (days), systemic anti-cytokine therapy given, time to first ICU admission (days), duration of ICU stay (days), highest temperature of fever, hypotension that required intervention, hypoxia that required supplemental oxygen, any other symptoms and whether patient dialyzed will be presented.

Listing of CRS information will be provided.

#### 8.15.1.2 ICANS AEs (Protocol amendment 8 onwards)

Listing of ICANS information will be provided.

## 8.15.1.3 Neurotoxicity AEs (Protocol amendments 1-7)

Similar summaries as the summary for TEAEs by SOC and PT will be presented also for neurotoxicity TEAEs. Data will also be listed.

#### 8.15.2 Clinical Laboratory Evaluations

Laboratory results for all haematology, coagulation and biochemistry (including serum ferritin) parameters will be listed in separate listings.

In addition, infectious disease screen results will be presented in a listing.

A listing containing the pregnancy test results will also be presented.

## 8.15.3 12-lead Electrocardiogram (ECG)

ECG will be performed during screening and at pre-conditioning phase (Day -6) and will be repeated if clinically indicated. The heart rate, PR, RR, QT intervals, QRS duration, corrected QT intervals and an overall interpretation will be collected.

All ECG assessment measurements will be listed.

## 8.15.4 Echocardiogram (ECHO) or Multiple Gated Acquisition (MUGA)

ECHO or MUGA will be performed during screening and will be repeated if patient experiences

Template Author: Version 5.0 25Jun2020



Final 1.0/ 21-Dec-2023

CRS or if clinically indicated. Generally, for a patient, the same procedure method (ECHO or MUGA) should be used throughout the study to allow for direct comparisons. The ECHO and MUGA will include an evaluation for left ventricular ejection fraction (LVEF).

All LVEF results from ECHO and MUGA assessment results will be listed.

## 8.15.5 Vital Signs

Temperature, systolic and diastolic blood pressure, pulse/heart rate, respiratory rate and oxygen saturation will be recorded. Blood pressure and pulse/heart rate measurements should be recorded with the patient in a seated position or supine. On Day 1, vital signs will be recorded immediately prior to AUTO3 infusion and every 30 mins (± 10 mins) for 4 hours post AUTO3 infusion, but no less than once a day.

All vital signs measurements will be listed.

## 8.15.6 Physical and Neurological Examination

A complete physical examination will be conducted at screening including a complete neurological examination. Also, physical and neurological examination will be conducted at subsequent visits during treatment and follow-up phases. Any detected abnormalities will be recorded as medical history (abnormalities noted before AUTO3 infusion) or adverse events (abnormalities noted after AUTO3 infusion) and will be summarized and listed as described in section 8.4 or section 8.15.1, respectively. No separate listing of physical and neurological examination data will be considered.

#### 8.15.7 Eastern Cooperative Oncology Group (ECOG) Performance Status

All ECOG performance assessments will be listed.

#### 8.15.8 Death information

The number and percentage of deaths and the primary reason for death, within 30 days and anytime post infusion will be presented on the Safety set.

Template Author: Version 5.0 25Jun2020



Final 1.0/ 21-Dec-2023

All patients who died and their reason for death will also be listed.

#### 8.15.9 Hospitalisation information

Listings of hospitalisation information and health encounters will be provided.

## 8.15.10 Subsequent therapies

Anti-cancer medications and therapies received post AUTO3 infusion will be listed.

## 9 Interim Analyses

Given the premature termination of the study, the interim analyses initially planned will not be performed.

# 10 Development safety update report

A development safety update report (DSUR) will include safety data. DSUR is intended to serve as an annual report to regulatory authorities at the DSUR anniversary of the study. DSUR anniversary is the date of first authorization anywhere in the world. DSUR shells will be created in a separate document.

## 11 Changes to Planned Analyses

The following are changes to the planned analyses from that stated in the protocol (Version 10.0):

- See section 6.1 Termination of the study based on this, the planned Interim analyses and Phase II analyses in the protocol will not be performed.
- Censoring of patients receiving a new anti-cancer treatment will be applied for the analysis of progression-free survival, in addition of the other censoring rules.
- Enrolled set is not being defined or used in the planned analysis.
- Efficacy analysis set is not being defined or used in the planned analysis. Instead,



Final 1.0/21-Dec-2023

evaluable set will be used for all the efficacy analyses.

- Decisions following SEC8 meeting (CMED delivery 20200129\_SEC9)
  - Declare 150x10^6 to 450x10^6 AUTO3 Regimen B as the recommended Phase 2 doses/range
  - o 900x10^6 (Regimen A): Will not open, no longer applicable.
  - o 900x10^6 (Regimen B): Will not open, no longer applicable
  - RP2D Cohort: All subjects after SEC9 meeting (planned Cmed delivery SEC10) when RP2D were declared
  - RP2D Outpatient Cohort: To be introduced in the up-coming Protocol Amendment 9

## 12 Document History

| Date | Version | Modified by | Brief details of changes made to template |
|---|---|---|---|
| 21Dec2023 | 1.0 | | Initial final version of SAP |

## 13 References

- [1] Simon R. (1989) Optimal two-stage designs for phase II clinical trials. <u>Control Clin Trials</u> 10(1):1-10.
- [2] Skolnik JM, Barrett JS, Jayaraman B, Patel D, Adamson PC. (2008) Shortening the timeline of pediatric phase I trials: the rolling six design. <u>J Clin Oncol</u> 26(2):190-5.
- [3] (CTCAE v4)

http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE 4.03 2010-06-14 QuickReference 5x7.pdf

[4] Cheson, BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, et al. (2014). Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol **32**(27):3059-3068.



Protocol: AUTO3-DB1

Statistical Analysis Plan: Final 1.0/21-Dec-2023

# 14 Appendices

## 14.1 APPENDIX A – Study assessments

Below schedules of assessments can be found in Protocol v10:

- Assessments from Screening to End of Treatment Phase
- Efficacy and Safety Follow-up
- Safety and Survival Follow-up

## 14.2 APPENDIX B – Lugano Classification (Cheson et.al 2014)

Patients with NHL will be evaluated using response criteria for Non-Hodgkin Lymphoma for Documenting Disease Response.

| Response | Site | PET-CT-Based Response | CT-Based Response |
|----------|------|-----------------------|------------------------------|
| Complete | | Complete | Complete radiologic response |
| | | | (all of the following) |

 BMSOP111/F2



Protocol: AUTO3-DB1

Statistical Analysis Plan: Final 1.0/21-Dec-2023

| | Non-measured lesion Organ | Not applicable Not applicable | Absent Regress to normal |
|---|---|---|---|
| | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | Regress to normal |
| | New lesions | None | None |
| | Bone marrow | No evidence of FDG-avid disease in marrow | Normal by morphology; if indeterminate, IHC negative |
| Partial | | Partial metabolic response | Partial remission (all of the following) |



Protocol: AUTO3-DB1

Statistical Analysis Plan: Final 1.0/21-Dec-2023

| | Lymph nodes<br>and<br>extralymphatic<br>sites | Score 4 or 5b with reduced uptake compared with baseline and residual mass(es) of any size. At interim, these findings suggest responding disease. At end of treatment, these findings indicate residual disease. | ≥50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of up to 6 target measurable nodes and extranodal sites. When a lesion is too small to measure on CT, assign 5 mm × 5 mm as the default value. When no longer visible, 0 × 0 mm For a node >5 mm × 5 mm, but smaller than normal, use actual measurement for calculation. |
|---|---|---|---|
| | Non-measured lesion | Not applicable | Absent/normal, regressed, but no increase |
| | Organ<br>enlargement | Not applicable | Spleen must have regressed by >50% in length beyond normal |
| | New lesions | None | None |
| | Bone Marrow | Residual uptake higher than uptake in normal marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed). If there are persistent focal changes in the marrow in the context of a nodal response, consideration should be given to further evaluation with MRI or biopsy or an interval scan. | Not applicable |
| No response or | | No metabolic response | Stable disease |



Protocol: AUTO3-DB1

Statistical Analysis Plan: Final 1.0/21-Dec-2023

| stable disease | | | |
|---|---|---|---|
| | Lymph nodes | Score 4 or 5 with no significant change in FDG | <50% decrease from baseline in SPD of up to 6 |
| | and | uptake from baseline at interim or end of | dominant, measurable |
| | extralymphatic | treatment | nodes and extranodal sites; no criteria for progressive |
| | sites | | disease are met. |
| | Non-measured | Not applicable | No increase consistent with progression |
| | lesion | | |
| | Organ | Not applicable | No increase consistent with progression |
| | enlargement | | |
| | New lesions | None | None |
| | Bone marrow | No change from baseline | Not applicable |
| Progressive | | Progressive metabolic disease | Progressive disease requires at least 1 of the following: |
| disease | | | |
| | Individual | Score 4 or 5 with an increase in intensity of | Cross product of the LDi and perpendicular diameter |
| | target | uptake | (PPD) progression |
| | nodes/nodal | from baseline and/or | (as defined below for extranodal lesions). |
| | masses | | |
| | Extranodal | New FDG-avid foci consistent with lymphoma | An individual node/lesion must be abnormal with: |
| | lesions | at interim or end-of-treatment assessment | LDi >1.5 cm, and increase by ≥50% from PPD nadir, and |
| | | | an increase in LDi or SDi from nadir: |
| | | | 0.5 cm for lesions ≤2 cm |
| | | | 1.0 cm for lesions >2 cm |
| | | | In the setting of splenomegaly, the splenic length must |
| | | | increase by >50% of the extent of its prior increase |
| | | | beyond baseline (e.g. a 15 cm spleen must increase to |
| | | | >16 cm). If no prior splenomegaly, must increase by at |
| | | | least 2 cm from baseline. |
| | | | New or recurrent splenomegaly |
| | Non-measured | None | New or clear progression of pre-existing non-measured |

 BMSOP111/F2



Protocol: AUTO3-DB1

Statistical Analysis Plan: Final 1.0/21-Dec-2023

| lesions | | lesions |
|---|---|---|
| New lesions | New FDG-avid foci consistent with lymphoma rather than another aetiology (e.g. infection, inflammation). If uncertain regarding aetiology of new lesions, biopsy or interval scan may be | Regrowth of previously resolved lesions A new node >1.5 cm in any axis. A new extranodal site >1.0 cm in any axis; if <1.0 cm in any axis, itspresence must be unequivocal and must be attributable to lymphoma Assessable disease of any size unequivocally attributable |
| | considered | to lymphoma |
| Bone marrow | New or recurrent FDG-avid foci | New or recurrent involvement |

5PS=5-point scale; CT=computed tomography; FDG=fluorodeoxyglucose; IHC=immunohistochemistry; LDi=longest transverse diameter of a lesion; MRI=magnetic resonance imaging; PET=positron emission tomography; PPD=cross product of the LDi and perpendicular diameter; SDi=shortest axis perpendicular to the LDi; SPD=sum of the product of the perpendicular diameters for multiple lesions.

- A score of 3 in many subjects indicates a good prognosis with standard treatment, especially if at the time of an interim scan. However, in trials involving PET where de-escalation is investigated, it may be preferable to consider a score of 3 as inadequate response (to avoid undertreatment). Measured dominant lesions: Up to 6 of the largest dominant nodes, nodal masses, and extranodal lesions selected to be clearly measurable in 2 diameters. Nodes should preferably be from disparate regions of the body and should include, where applicable, mediastinal and retroperitoneal areas. Non-nodal lesions include those in solid organs (e.g. liver, spleen, kidneys, lungs), GI involvement, cutaneous lesions, or those noted on palpation.
  - Non-measured lesions: Any disease not selected as measured, dominant disease and truly assessable disease should be considered not measured. These sites include any nodes, nodal masses, and extranodal sites not selected as dominant or measurable or that do not meet the requirements for measurability, but are still considered abnormal, as well as truly assessable disease, which is any site of suspected disease that would be difficult to follow quantitatively with measurement, including pleural effusions, ascites, bone lesions, leptomeningeal disease, abdominal masses, and other lesions that cannot be confirmed and followed by imaging. In Waldeyer's ring or in extranodal sites (e.g. GI tract, liver, bone marrow), fluorodeoxyglucose uptake may be greater than in the mediastinum with complete metabolic response, but should be no higher than surrounding normal physiologic uptake (e.g. with marrow activation as a result of chemotherapy or myeloid growth factors).
- PET 5PS: 1, no uptake above background; 2, uptake ≤mediastinum; 3, uptake >mediastinum but ≤liver; 4, uptake moderately >liver; 5, uptake markedly higher than liver and/or new lesions; X, new areas of uptake unlikely to be related to lymphoma

 BMSOP111/F2



Protocol: AUTO3-DB1

**Statistical Analysis Plan:** 

Final 1.0/ 21-Dec-2023

## 14.3 APPENDIX C – Clinical Laboratory Tests Performed by Local Laboratory

| Description |
|---|
| Haemoglobin, red blood cell count, platelet count, white blood cell (WBC)count with differential (neutrophils, eosinophils, lymphocytes, monocytes, and basophils). |
| Prothrombin time, international normalised ratio, activated partial thromboplastin time, fibrinogen. |
| Sodium, phosphate, potassium, alanine aminotransferase (ALT), aspartate aminotransferase (AST), uric acid, urea, creatinine, creatine phosphokinase (CPK), lactate dehydrogenase, total bilirubin, calcium, albumin. All tests must be performed prior to AUTO3 infusion on Day 0. |
| Ferritin, C-reactive protein. |
| Serum ( $\beta$ -human chorionic gonadotropin) or urine pregnancy testing for females of childbearing potential. |
| <ul> <li>HIV antibody.</li> <li>Hepatitis B core antibody: if positive, further testing (deoxyribonucleic acid [DNA] by PCR) to rule out active disease or chronic carrier. Must be confirmed negative prior to screening.</li> <li>Hepatitis C virus antibody: if positive for hepatitis C virus, further testing (by ribonucleic acid PCR) should be performed to rule out active infection.</li> <li>Anti-HTLV-1.</li> <li>Anti-HTLV-2.</li> <li>Syphilis Serology.</li> </ul> |

DNA = deoxyribonucleic acid; HIV = human immunodeficiency virus; HTLV = human T-cell lymphocyte virus; PCR = polymerase chain reaction.



Protocol: AUTO3-DB1

Statistical Analysis Plan:

Final 1.0/ 21-Dec-2023

## 14.4 Tables, Figures and Listing shells

A separate document was considered to cover the tables, figures and listings shells.

# **DocuSign**

## **Certificate Of Completion**

Envelope Id: F01779750CED428BB52119A922B04034

Subject: Complete with DocuSign: AUTO3-DB1\_SAP\_Final v1.0.doc

Source Envelope:

Document Pages: 49 Certificate Pages: 5 Signatures: 3 Initials: 0

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Status: Completed

Envelope Originator:



Sent: 08-Jan-2024 | 12:49 Viewed: 08-Jan-2024 | 12:49 Signed: 08-Jan-2024 | 12:50

#### Record Tracking

Status: Original

(Required)

08-Jan-2024 | 12:46

Holder:

Location: DocuSign

**Timestamp** 

## Signer Events

Cmed (Clinical Research Services) Limited Security Level: Email, Account Authentication (Required) Signature

Signature Adoption: Pre-selected Style Signature ID:

1BBA474B-F893-46E8-823C-A9A72C9ACC9B

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I am the author of this document

**Electronic Record and Signature Disclosure:** 

Accepted: 08-Jan-2024 | 12:49

Security Level: Email, Account Authentication

ID: b62a27d0-69eb-4542-895d-69922330f025

Signature Adoption: Pre-selected Style Signature ID:

A3C726D3-5BE9-4A51-84EB-20EF132C7965

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

Ich genehmige dieses Dokument

Electronic Record and Signature Disclosure: Accepted: 08-Jan-2024 | 12:51

ID: e4a707d8-bd8c-4fc6-b8b5-f4ad129a037d

Sent: 08-Jan-2024 | 12:49 Viewed: 08-Jan-2024 | 12:51 Signed: 08-Jan-2024 | 12:52

# Signer Events

Security Level: Email, Account Authentication (Required), Login with SSO

## **Signature**

## **Timestamp**

Sent: 08-Jan-2024 | 12:49 Viewed: 08-Jan-2024 | 19:05 Signed: 08-Jan-2024 | 19:14

Signature Adoption: Pre-selected Style Signature ID:

3D469D59-6D48-4F9A-BA53-CDD0E6D56E5B

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

#### Electronic Record and Signature Disclosure:

Accepted: 08-Jan-2024 | 19:05 ID: 188d99b5-c246-46ef-915c-2530f381b6b6

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 08-Jan-2024 12:49<br>08-Jan-2024 19:05<br>08-Jan-2024 19:14<br>08-Jan-2024 19:14 |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Cmed (Clinical Research Services) Limited (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

## Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

## How to contact Cmed (Clinical Research Services) Limited:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: dataprivacy@cmedresearch.com

## To advise Cmed (Clinical Research Services) Limited of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at dataprivacy@cmedresearch.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

## To request paper copies from Cmed (Clinical Research Services) Limited

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to dataprivacy@cmedresearch.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

## To withdraw your consent with Cmed (Clinical Research Services) Limited

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to dataprivacy@cmedresearch.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

## Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

## Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Cmed (Clinical Research Services) Limited as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Cmed (Clinical Research Services) Limited during the course of your relationship with Cmed (Clinical Research Services) Limited.